CLINICAL TRIAL: NCT02342535
Title: Community-Clinic Partnership to Promote Physical Activity in South Asian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Metropolitan Asian Family Services (Unknown)
Responsible Party: Principal Investigator, Namratha Kandula, Assitant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU00101433
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical activity intervention (Other): Participants will attend bi weekly exercise classes for a total of 16 weeks, led by certified, and trained instructors.
  The participant's children between the ages of 6 and 14 years will participate in the martial arts class with the mothers.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Culturally tailored physical activity intervention for South Asian women and their children.

SUMMARY:
The goal of this study is to pilot-test a culturally-salient physical activity intervention, using a randomized design, among under served, overweight/obese South Asian women at high risk for developing Diabetes.

DETAILED DESCRIPTION:
Regular physical activity prevents type 2 diabetes mellitus (DM). Although physical inactivity and DM are common in the United States (US), the investigators data, and others,have shown that Asian Indian and Pakistani (South Asian) women are at even greater risk. South Asians (SA) are one of the fastest growing segments of the US population.Studies show that SA women have a markedly higher DM prevalence and are less physically active than women from other racial/ethnic groups.SA also have greater insulin resistance and visceral adiposity at a lower body mass index (BMI). A combination of regular, moderate intensity physical activity (PA) and resistance exercises has been shown to decrease visceral adiposity and improve insulin sensitivity, even without weight loss; thus, PA may be especially important for DM prevention among SA women. Despite being at increased risk, very few evidence-based DM prevention and PA interventions exist for SA women in the US.

This proposal builds on a successful academic-community partnership between Northwestern University and Metropolitan Asian Family Services, an organization that provides health care and social services to lower-income SA immigrant families. The partnership has focused on translating and implementing evidence-based lifestyle interventions for SA immigrants in real-world, clinic and community settings. The investigators formative research found that SA women, in particular, were not being reached by current efforts to promote PA. Importantly, however, the main reasons for the reduced effectiveness of traditional strategies for PA promotion related more to socio-cultural perceptions and beliefs than simply to language barriers. SA women reported little PA and had difficulty even defining exercise. Although 75% of women were sedentary and overweight, they did not recognize these as risk factors for DM. Lack of knowledge about benefits of PA, cultural and linguistic isolation, concerns about modesty, and rigid gender roles strongly influenced SA women's proclivity for physical inactivity. In this context, much more work will be needed to address SA women's physical inactivity than simple language translation of proven lifestyle interventions.

ELIGIBILITY:
Inclusion Criteria:

* Should meet all the 3 criteria below and meet the criteria for option 4 below or should meet the criteria for 5 as well as 6.

  1. Self-identified as South Asian
  2. Women
  3. Have children between the ages of 6 and 14 years. AND Meet either of the criteria below
  4. History of gestational diabetes during any of the pregnancies Or
  5. Body Mass Index between 25 and 35 kg/m2 And
  6. Family history of diabetes in a first degree relative.

Exclusion Criteria:

* Blood pressure of over 160/100 mm Hg
* History of diabetes
* Saying Yes to any question on the Exercise Assessment and Screening for You (EASY) exercise screening tool
* Currently pregnant or trying to get pregnant in the next year
* Planning to move out of Illinois in the next 6 months.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Namratha Kandula, MD,MPH, Principal Investigator — Assistant Professor, Northwestern University
Locations (2):
- United States (2):
  - Northwestern University-Feinberg School of Medicine, Chicago, Illinois
  - Metropolitan Asian Family Services, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total number of participants who signed up for the study were 68 and not 71.
Groups:
- Physical Activity Intervention: Participants will attend bi weekly exercise classes for a total of 16 weeks, led by certified, and trained instructors.
  The participant's children between the ages of 6 and 14 years will participate in the martial arts class with the mothers.
  Physical Activity: Culturally tailored physical activity intervention for South Asian women and their children.
Period: Overall Study
Arm/Group | Physical Activity Intervention
Started | 68 (30 women who participated in the aerobic exercise class and 38 children.)
Completed | 68 (30 women in aerobic class and 38 kids in kids exercise class)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 30 South Asian adult women were the participants whose data is being analyzed. No research data was obtained from the children. The children have only assented to be in the study.
Groups:
- Physical Activity Intervention: Participants will attend bi weekly exercise classes for a total of 16 weeks, led by certified, and trained instructors.
  The participant's children between the ages of 6 and 14 years will participate in the martial arts and yoga class with their mothers.
  Physical Activity: Culturally tailored physical activity intervention for South Asian women and their children.
Arm/Group | Physical Activity Intervention
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants were enrolled into the study from November 2014 to February 2015. The average age of mothers was 40 (SD±5) years.
  years | 40 (5)
Sex/Gender, Customized [Number; unit: participants]
  Female Parent | 30
  Female Child | 17
  Male Child | 21
Race/Ethnicity, Customized [Number; unit: participants]
  South Asian | 68
Region of Enrollment [Number; unit: participants] — Majority participants from the Rogers Park neighborhood of Chicago and the neighboring suburbs in Illinois.
  participants
    United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity (Minutes/Week)
Description: To test for differences in physical activity, we used mixed-effects models for pre- and post-intervention accelerometer data. In these models, the outcome was daily minutes of bout corrected moderate-vigourous physical activity. Time (pre/post-intervention) was treated as a binary variable in order to measure changes in physical activity. Models controlled for accelerometer wear time and weekend day.
Time Frame: Baseline and 4 months
Population: We did not collect any data from the children, so all the data analysis is from the data obtained from the 30 mothers. To test for differences in physical activity, we used mixed-effects models for pre- and post-intervention accelerometer data. In these models, the outcome was daily minutes of bout corrected moderate-vigourous physical activity.
Measure: Mean (Standard Deviation); unit: minute/week activity
Groups:
- Physical Activity Intervention: Participants will attend bi weekly exercise classes for a total of 16 weeks, led by certified, and trained instructors.
  The participant's children between the ages of 6 and 14 years will participate in the kids exercise class with their mothers.
  Physical Activity: Culturally tailored physical activity intervention for South Asian women and their children.
Arm/Group | Physical Activity Intervention
Number analyzed (Participants) | 30
minute/week activity
  Baseline | 42 (104)
  Post intervention at 4 months | 58 (117)

ADVERSE EVENTS:
Arm/Group | Physical Activity Intervention
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 0/68

LIMITATIONS AND CAVEATS:
Limitations of this pilot study are inclusion of a single site in Chicago, lack of a control arm, and that we were only able to recruit and enroll 20% of the individuals we approached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No